CLINICAL TRIAL: NCT05040464
Title: Comparison of Azathioprine to Methotrexate in Combination Therapy With Adalimumab in Crohn's Disease: an Open-label Randomized Controlled Trial
Acronym: COMET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Nantes University Hospital (Other); AP-HP - HU BEAUJON (Unknown); CHU REIMS (Unknown); Centre Hospitalier Universitaire de Besancon (Other); CHRU LILLE (Unknown); University Hospital, Bordeaux (Other); Henri Mondor University Hospital (Other); Hospices Civils de Lyon (Other); CHU Rennes,France (Unknown); CHU ROUEN - HOPITAL DE BOIS-GUILLAUME (Unknown); CHRU TOURS (Unknown); University Hospital, Toulouse (Other); University Hospital, Montpellier (Other); CHU NICE (Unknown); CHU NANCY (Unknown); CHU CAEN (Unknown); CHU SAINT-ETIENNE (Unknown); CH TOURCOING (Unknown); Hopitaux Civils de Colmar (Other); CH COTE BASQUE (Unknown); CH ROUBAIX (Unknown); CHI CRETEIL (Unknown); CHI TOULON LA SEYNE (Unknown); CH VALENCE (Unknown); CMC Ambroise Paré, Pierre Cherest, Hartmann (Unknown); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0080
Record Dates: First submitted 2021-08-26; First posted 2021-09-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Azathioprine; Methotrexate
Keywords: Crohn Disease; Combinations of therapy; anti-Tumor Necrosis Factor; azathioprine; methotrexate
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZA group (Experimental): Combination of sub-cutaneous administration of adalimumab at a dose of 160mg(W0)-80mg(W2)-40mg(W6) and then 40mg EOW and oral AZA capsules at a daily dose of 2.5 mg/kg
  Interventions: Drug: AZA capsules; Biological: blood sample
- MTX group (Experimental): Combination of sub-cutaneous administration of adalimumab at a dose of 160mg (week (W) 0)-80mg(W2)-40mg(W6) and then 40mg EOW and sub-cutaneous MTX 25mg once a week
  Interventions: Drug: MTX; Biological: blood sample

INTERVENTIONS:
Drug: AZA capsules — oral AZA capsules at a daily dose of 2.5 mg per kilogram,
  Arms: AZA group
Drug: MTX — MTX 25 mg SC once a week
  Arms: MTX group
Biological: blood sample — The lab tests are: serum albumin, C-reactive protein, thrombocytosis and haemoglobin.

SUMMARY:
Combination therapy, the association of an anti-Tumor Necrosis Factor (TNF) to an immunosuppressant, is recognized as the most effective treatment during Crohn's disease (CD). Several mechanisms have been proposed to explain the superiority of combination therapy over monotherapy, the additive effect of two effective drugs or the prevention of anti-TNF immunogenicity. As the best combination therapy is unknown, both azathioprine (AZA) and methotrexate (MTX) are used. Some retrospective studies suggest a higher effectiveness of AZA. MTX may have an advantage in terms of safety.

The investigators hypothesize that AZA is more effective than MTX as combination therapy with adalimumab to improve short-term endoscopic, clinical and pharmacological outcomes in CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with age > 18 years
* Crohn's disease for at least 6 weeks,
* Clinically active with CDAI > 150
* Active inflammation by endoscopy (CDEIS > 4) at baseline
* Not responder to conventional therapy or are intolerant to or have medical contraindications for such therapies and initiating treatment with adalimumab
* Patient followed in a center belonging to the GETAID network
* Fertile men and women of childbearing potential included in the protocol should use adequate methods of contraception according to study drug SMPCs.
* Written consent

Exclusion Criteria:

* Short bowel syndrome, ostomy, symptomatic stricture, abscess, recent history of abdominal surgery (<3 months)
* Non-passable colonic stricture
* Previous intolerance to thiopurines or MTX
* Previous exposition to adalimumab
* Contra-indication to immunosuppressants or anti-TNF
* Others serious simultaneous illness that could interfere with study participation
* Planning pregnancy, pregnancy or lactation or absence of contraception
* Known substance abusers
* Use of any investigational drug within 30 days
* Adults protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Variation of the endoscopic response between AZA and MTX groups | 26 weeks
  Variation of the endoscopic response to AZA in combination with adalimumab and to MTX in combination with adalimumab in patients with CD.
  The endoscopic reference score (EREFS) is used to determine severity of 5 endoscopic findings: edema, rings, exudates, furrows, and structures. The EREFS classification system rates the severity of edema (0-2), rings (0-3), exudates (0-2), furrows (0-2), and strictures (0-1)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No